CLINICAL TRIAL: NCT03330379
Title: Comparison of Two Strategies for the Prevention of Endotracheal Tube Cuff Underinflation During Invasive Mechanical Ventilation: Intermittent Versus Continuous Cuff Pressure Control - A Randomised Controlled Study
Brief Title: Comparison of Two Strategies for Endotracheal Tube Cuff Underinflation Prevention During Invasive Mechanical Ventilation
Acronym: CONTIPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC16_0390
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Acute Brain Injury; Brain Injuries
Keywords: Endotracheal tube; ventilator's associated pneumonia; intensive care unit; orotracheal intubation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuous adjustment strategy (Experimental): patients assigned to the continuous adjustment strategy, in addition to standard care, the Tracoe Smart CuffmanagerTM will be connected to the tracheal cuff
  Interventions: Device: Tracoe Smart CuffmanagerTM
- usual care (No Intervention): patients with usual care

INTERVENTIONS:
Device: Tracoe Smart CuffmanagerTM — In patients randomly assigned to the continuous adjustment strategy, in addition to standard care, the Tracoe Smart CuffmanagerTM will be connected to the tracheal cuff. Within the 2 days following the inclusion, all the intermittent Pcuff measurements will be collected as well as the incidence of Pcuff manual adjustments
  Arms: continuous adjustment strategy

SUMMARY:
During invasive mechanical ventilation, maintaining endotracheal tube cuff pressure (Pcuff) around 25 cmH2O is recommended for sealing the upper airways. The continuous control of Pcuff with a simple mechanical device, the Tracoe Smart CuffmanagerTM, has never been assessed. The investigators hypothesize that the Tracoe Smart CuffmanagerTM would allow a reduction of the incidence of underinflation episodes, as compared with the intermittent strategy of Pcuff control.

DETAILED DESCRIPTION:
During invasive mechanical ventilation, maintaining a tracheal cuff pressure (Pcuff) around 25 cmH2O is recommended to prevent cuff over- (> 30 cmH2O) and underinflation (< 20 cmH2O), identified as risk factors for tracheal ischemic damage and for oropharyngeal microaspirations, respectively. Intermittent measurements with intermittent adjustments of Pcuff is the widely used strategy but, between measurements, over- and underinflation episodes could occur. Devices allowing a continuous control of Pcuff are therefore appealing. As microaspiration is the most relevant mechanism for ventilator-associated pneumonia (VAP), the use of such devices may decrease the incidence of VAP for instance. To the knowledge of the investigators, the continuous control of Pcuff with a simple mechanical device, the Tracoe Smart CuffmanagerTM, has never been assessed. The investigators hypothesize that the Tracoe Smart CuffmanagerTM would allow a reduction of the incidence of underinflation episodes, as compared with the intermittent strategy of Pcuff control. As secondary objectives, the investigators aim to assess the impact of the use of the Tracoe Smart CuffmanagerTM on the incidence of overinflation episodes and on the incidence of early ventilator-associated pneumonia. A homogenous population will be studied for this purpose: patients admitted with severe acute brain damage.

ELIGIBILITY:
Inclusion Criteria:

* with severe acute brain damage
* admitted in the ICU for less than 48 hours
* and expected to receive invasive mechanical ventilation (through orotracheal tube with a low pressure-high volume cuff) for at least 48 hours after inclusion.

Exclusion Criteria:

* change in the upper airway management within the 48 hours following the inclusion (extubation or change in the tracheal tube or tracheostomy)
* pregnancy, moribund status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of underinflation episodes | Day2
  The primary outcome is to test whether the Tracoe Smart CuffmanagerTM reduces the incidence of underinflation episodes, as compared with the intermittent strategy of Pcuff control. Therefore, a comparison, between the 2 groups, of the incidence of Pcuff <20 cmH2O measurements will be performed.
  Time Frame: Within the 2 days following the inclusion, all the intermittent Pcuff measurements will be collected as well as the incidence of Pcuff manual adjustments

SECONDARY OUTCOMES:
incidence of Pcuff >30 cmH2O measurements (overinflation episodes) | Within the 2 days following the inclusion
  As secondary objective, a comparison, between the 2 groups, of the incidence of Pcuff >30 cmH2O measurements (overinflation episodes) will be performed.
  Furthermore, the incidence of early ventilator-associated pneumonia will be compared between the 2 groups.
Duration of mechanical ventilation | Within the 2 days following the inclusion
ICU length of stay | Within the 2 days following the inclusion
ICU mortality | Within the 2 days following the inclusion
occurrence of early ventilator-associated pneumonia | During the first two weeks of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Dauvergne, Principal Investigator — Nantes University Hospital
Locations (1):
- Chu de Nantes, Nantes, France

REFERENCES:
- [Derived] Dauvergne JE, Geffray AL, Asehnoune K, Rozec B, Lakhal K. Automatic regulation of the endotracheal tube cuff pressure with a portable elastomeric device. A randomised controlled study. Anaesth Crit Care Pain Med. 2020 Jun;39(3):435-441. doi: 10.1016/j.accpm.2020.04.007. Epub 2020 May 4. PMID 32376293